CLINICAL TRIAL: NCT01281332
Title: Evaluation of a Novel Mechanical Device for Relief of Menopausal Vasomotor Symptoms.
Brief Title: Mechanical Device for the Relief of Hot Flashes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Alexander Medical Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Robert Reid, Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OBGY-208-10
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Hot Flashes
Keywords: menopause; hot flash; quality of life
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menopod device (Active Comparator): Menopod®
  Interventions: Device: Menopod
- Sham device (Sham Comparator): Inactive device.
  Interventions: Device: Inactive device

INTERVENTIONS:
Device: Menopod — The mechanism of action of the device will not be revealed in advance.
  Arms: Menopod device
Device: Inactive device
  Other Names: The mechanism of action of the active device is disabled.
  Arms: Sham device

SUMMARY:
Hypothesis: A mechanical device when applied to the back of the neck at the onset of a menopausal hot flash will attenuate the severity and duration of symptoms providing women with a reassuring non-hormonal intervention to improve quality of life in the menopausal transition. This pilot study will evaluate the effectiveness of this unit.

The mechanism of action of the device will not be revealed in advance.

DETAILED DESCRIPTION:
This is a pilot study to test logistics and gather information for planning the definite trial. We will randomly allocate 40 subjects to receive either the active Menopod device (n=20) or a sham device with the mechanism disabled (n=20).

We will recruit menopausal women with moderate to severe hot flashes (as defined by FDA standards this means a minimum of 7 per day).

The two primary outcome parameters are the hot flash score which is the product of frequency x intensity (Sloan 2001), and the average duration (in minutes) of hot flash episodes over the course of one day. These outcomes will be self-recorded by subjects in a diary designed by our research team on five separate days throughout the course of the study, once during the evaluation phase and once per week over the four week treatment phase. The two summary measures will be the changes from baseline to the last record collected for hot flash scores and average durations. Delta values (assessment phase minus fourth treatment period) will be compared between the two treatment groups (active versus sham device) using t tests (IBM SPSS Statistics version 21).

ELIGIBILITY:
Inclusion Criteria:

* Age range: 40 to 65 years
* Healthy postmenopausal woman
* natural or surgical menopause
* FSH > 30 IU/L
* Amenorrhea > 6 months prior to study
* Minimum of 7 moderate hot flashes per day documented in diary during evaluation phase

Exclusion Criteria:

* Any therapy for hot flashes prior to or during study
* Obesity: BMI > 35
* Alcohol abuse
* Drug abuse
* Unable to use device as per protocol
* Unable to complete required documentation
* Serious medical condition:
* coronary heart disease
* stroke
* chronic renal or hepatic disease
* diabetes
* depression or other psychiatric illness
* cancer

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Hot flash score and duration | Change from baseline to end of study (week 4).
  Hot flash score is a product of frequency x intensity (Sloan 2001). Duration (minutes) will be recorded in diary.

SECONDARY OUTCOMES:
Quality of Life (QOL) and Anxiety | Change from baseline to end of study (week 4).
  Subjects will complete the Hot Flash Related Daily Interference Scale once during the evaluation phase and once per week over the four week treatment phase (Carpenter 2001). This validated questionnaire assesses the impact of hot flashes on daily activities and overall QOL. They will also complete the Zung Self-Rating Anxiety Scale (Zung 1971). This validated 20-item questionnaire measures anxiety with established normal, mild to moderate, marked to severe and extreme levels.
  Carpenter JS. The Hot Flash Related Daily Interference Scale: a tool for assessing the impact of hot flashes on quality of life following breast cancer. J Pain Symptom Manage 2001 Dec;22(6):979-89.
  Zung WW. A rating instrument for anxiety disorders. Psychosomatics 1971 Nov-Dec;12(6):371-9.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Reid, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Background] Sloan JA, Loprinzi CL, Novotny PJ, Barton DL, Lavasseur BI, Windschitl H. Methodologic lessons learned from hot flash studies. J Clin Oncol. 2001 Dec 1;19(23):4280-90. doi: 10.1200/JCO.2001.19.23.4280. PMID 11731510
- [Background] Carpenter JS. The Hot Flash Related Daily Interference Scale: a tool for assessing the impact of hot flashes on quality of life following breast cancer. J Pain Symptom Manage. 2001 Dec;22(6):979-89. doi: 10.1016/s0885-3924(01)00353-0. PMID 11738160
- [Background] Zung WW. A rating instrument for anxiety disorders. Psychosomatics. 1971 Nov-Dec;12(6):371-9. doi: 10.1016/S0033-3182(71)71479-0. No abstract available. PMID 5172928